CLINICAL TRIAL: NCT06868485
Title: A Phase II, Open Label, Multicenter, Single Arm Study of WSD0922-FU for Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer With First-Line Osimertinib Treatment and Harbor a C797S Mutation
Brief Title: A Study to Assess the Efficacy of WSD0922-FU in Patients With C797S+ Advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wayshine Biopharm, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WS2202
Record Dates: First submitted 2025-02-22; First posted 2025-03-11 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: C797S; BM; WSD0922-FU; NSCLC; EGFR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose level A selected from Phase I study (Experimental): BID
  Interventions: Drug: WSD0922-FU Tablets, Dose level A
- Dose level B selected from Phase I study (Experimental): BID
  Interventions: Drug: WSD0922-FU Tablets, Dose level B

INTERVENTIONS:
Drug: WSD0922-FU Tablets, Dose level A — Oral, 21 days in each cycle
  Other Names: WSD0922
  Arms: Dose level A selected from Phase I study
Drug: WSD0922-FU Tablets, Dose level B — Oral, 21 days in each cycle
  Other Names: WSD0922
  Arms: Dose level B selected from Phase I study

SUMMARY:
This is a Phase II, Open Label, Multicenter, Single Arm Study of WSD0922-FU for Patients with Locally Advanced or Metastatic Non-Small Cell Lung Cancer whose Disease has Progressed with First-Line Osimertinib Treatment and whose Tumors harbor a C797S mutation within the Epidermal Growth Factor Receptor Gene.

DETAILED DESCRIPTION:
WSD0922-FU is a potent reversible inhibitor of both the single EGFRm+ (TKI sensitivity conferring mutation) and dual EGFRm+/C797S+ (third-generation TKI as first-line resistance conferring mutation) receptor forms of EGFR with selectivity margin over wild-type EGFR. Therefore WSD0922-FU has the potential to provide clinical benefit to patients with advanced NSCLC harboring both the single sensitivity mutations and the resistance mutation following first-line therapy with a third-generation EGFR TKI (e.g., Osimertinib). The clinical development program with WSD0922-FU will assess the safety and efficacy of WSD0922-FU in patients with advanced NSCLC whose cancers have progressed with or without brain metastasis following a first-line Osimertinib treatment.

ELIGIBILITY:
Inclusion criteria:

* Provision of signed and dated, written informed consent prior to any study-specific procedures, sampling and analyses.
* Male or female aged ≥18 years old.
* Histological or cytological confirmation diagnosis of NSCLC.
* Locally advanced or metastatic NSCLC, not amenable to curative surgery or radiotherapy.
* Evidence of radiological disease progression while on a previous continuous treatment with first-line Osimertinib treatment.
* Documented EGFR mutation .
* Eastern Cooperative Oncology Group (ECOG) 0-1 and a minimum life expectancy of 12 weeks.
* At least one lesion, not previously irradiated and not chosen for biopsy during the study.
* Females should have evidence of non-childbearing potential.

Exclusion criteria:

* Any investigational agents or other anticancer drugs from a previous treatment regimen or clinical study within 14 days of the first dose of study treatment.
* Any unresolved toxicities from prior therapy greater than CTCAE Grade 1.
* Symptomatic brain complications that require urgent neurosurgical or medical intervention.
* Any evidence of severe or uncontrolled systemic diseases.
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection.
* Past medical history of ILD.
* Inadequate bone marrow reserve or organ function as demonstrated.
* Males and females of reproductive potential.
* Known intracranial hemorrhage which is unrelated to tumor.
* Seizures requiring a change in anti-epileptic medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | every 8 weeks, up to 1 year
  proportion of patients with a best overall response of complete response or partial response

SECONDARY OUTCOMES:
Duration of Response (DoR) | every 8 weeks, up to 1 year
  proportion of patients with the time from the date of first documented response until the date of documented progression or death in the absence of disease progression
PFS | every 8 weeks, up to 1 year
  proportion of patients with the time from randomization until the date of objective disease progression or death
Disease Control Rate (DCR) | every 8 weeks, up to 1 year
  the percentage of patients who have a best overall response of CR or PR or SD
Overall Survival (OS) | 24 months
  the time from the date of randomization until death due to any cause
EORTC QLQ-C30 (HRQoL) | up to 24 months
  PROs will be assessed using the EORTC QLQ-C30,changes in score compared to baseline will be evaluated.
EORTC QLQ-LC13 (HRQoL) | up to 24 months
  PROs will be assessed using the EORTC QLQ-LC13, changes in score compared to baseline will be evaluated.
PRO CTCAE (HRQoL) | up to 24 months
  To be assessed using the PRO CTCAE ,changes in symptoms compared to baseline will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Adjei Alex A., PhD, Principal Investigator — The Cleveland Clinic
Locations (18):
- United States (8):
  - FOMAT Oncology, Oxnard, California
  - Cleveland Clinic Weston Hospital, Weston, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - Hackensack Meridian Health-Southern Ocean Medical Center, Manahawkin, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - TxO Central/South, Texas Oncology -Central/South Texas, Austin, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- China (5):
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Wuhan Union Hospital, Wuhan, Hubei
  - Shanghai East hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
- France (5):
  - Centre Hospitalier Universitaire (CHU) de Rennes - Hopital de Pontchaillou, Rennes, Ille-et-Vilaine
  - Centre Francois Baclesse, Caen, Normandy
  - Centre Hospitalier Universitaire CHU De Limoges, Limoges, Nouvelle-Aquitaine
  - CHU Bordeaux - Centre Francois Magendie, Pessac, Nouvelle-Aquitaine
  - CHU Toulon - Hopital Sainte Musse, Toulon, Var

IPD SHARING:
Plan to Share IPD: No